CLINICAL TRIAL: NCT03192540
Title: The Impact of an 8-week Supported Exercise Program on Fitness and Symptoms of Anxiety and Depression in Adolescents With Down Syndrome
Brief Title: The Impact of an 8-week Supported Exercise Program on Fitness and Symptoms in Adolescents With Down Syndrome
Acronym: DSFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Emily Jean Davidson, MD, MPH, Doctor, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P00023661
Record Dates: First submitted 2017-05-15; First posted 2017-06-20 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Down Syndrome
Keywords: Exercise; Fitness; Overall wellbeing
MeSH Terms: conditions — Down Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): These are participants who will be undergoing exercise intervention.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will undergo an exercise protocol once a week, for eight weeks. Exercise will be continuous for one hour.

SUMMARY:
This study explores the effects of an eight-week exercise intervention for adolescents with Down syndrome on home exercise compliance. As well, to observe changes in fitness including muscular strength, endurance and aerobic capacity. Finally to observe any changes in mood, behavior and quality of life.

DETAILED DESCRIPTION:
Adolescents with Down syndrome will participate in an eight-week, center-based exercise intervention. Participants will undergo an hour of exercise intervention each week. During this time, participants will be working with a team consisting of a physician, physical therapy student volunteers, and clinical research coordinators. Exercises will focus on strength and endurance of all major muscle groups, while ensuring proper technique and form is used. They will also receive instruction on how to continue the exercise program at home.

Prior to starting, and at the end of eight sessions, all exercise participants will undergo testing procedures for anthropometric, strength and flexibility measurements. This data will be collected as part of clinically evaluating the impact of the program on each participant. In addition to the exercise program (and clinical assessments of fitness), DSFit participants will complete study measures of behavioral functioning as well as scales of depression and anxiety. Participants in the DSFit study will also complete a weekly exercise log during the intervention and for a follow-up period afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 10 to 17 years old (until 18th birthday)
* Diagnosed with Down syndrome by a physician
* Medically cleared to exercise

Exclusion Criteria:

* Requires consistent one-on-one care
* History of behavioral issues (outbursts, aggressive/self-injurious, bolting)
* Pre-existing cardiovascular, respiratory or orthopedic conditions that could place participant at risk for injury or illness resulting from exercise. For example:
* Untreated significant atlantoaxial instability
* Severe pulmonary hypertension

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Home Exercise Compliance | 2 months post completion of the exercise program
  To establish if the participant is performing the same amount of exercise each week, for up to three months after the stopped visiting the group exercise sessions.

SECONDARY OUTCOMES:
Muscular strength & endurance | The test will be performed before the exercise intervention and then after 8 weeks of exercise intervention.
  Participants will perform body-weight exercises that focus on upper body, lower body, core, and flexibility.
Aerobic capacity | The test will be preformed before the exercise intervention and then after 8 weeks of exercise intervention.
  Participants will complete the 6 minute walk test, where the investigators will receive an estimate measure of maximum aerobic fitness. Investigators will also collect heart rate and blood pressure as pre and post measurements when possible.
Anxiety and Depression Symptoms | The scale will be given the before the exercise intervention begins and then after 8 weeks of exercise intervention.
  Patient-Reported Outcomes Measurement Information System (PROMIS) - Parent report questionnaires
Behavioral Symptoms | The scale will be given the before the exercise intervention begins and then after 8 weeks of exercise intervention.
  Vanderbilt Scale - parent report questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No